CLINICAL TRIAL: NCT02428426
Title: Mucosal Microbiome in Human Gastric Intestinal Metaplasia and Duodenal Tissue.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Mucosal Microbiome in human gastric Intestinal Metaplasia and duodenal tissue., Shandong University
Other Study IDs: 2015SDU-QILU-G04
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Mucosal Microbiome; Gastric Intestinal Metaplasia; Duodenum
Keywords: Mucosal Microbiome; gastric intestinal metaplasia; duodenum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The metagenome was obtained from biopsy specimen.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- gastric intestinal metaplasia: patients were diagnosed gastric intestinal metaplasia
  Interventions: Other: endomicroscopy, targeted biopsy and 16s rRNA gene sequencing
- gastritis: patients were diagnosed non atrophic gastritis
  Interventions: Other: endomicroscopy, targeted biopsy and 16s rRNA gene sequencing

INTERVENTIONS:
Other: endomicroscopy, targeted biopsy and 16s rRNA gene sequencing

SUMMARY:
To investigate the mucosal microbiome in human gastric intestinal etaplasia and duodenal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for gastroendoscopy examination Aged between 18 and 80 years old

Exclusion Criteria:

* Antibiotic, probiotic or prebiotic usage within 2months,gastric inhibitor usage within 1 month Esophageal, gastric or duodenal cancer or other malignancy History of upper GI tract surgery Coagulopathy or bleeding disorders Allergy to fluorescein sodium Pregnant or breast-feeding (for females) Impaired renal function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective patients scheduled for pCLE examination at Qilu Hospital, Shandong University
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
The operational taxonomy units in gastric Intestinal Metaplasia and and Duodenal mucosal microbiome | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: li yanqing, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China